CLINICAL TRIAL: NCT04486664
Title: Effect of Mediterranean Diet on Metabolic Parameters and Microbiome in Dyslipidemic Patients: Randomized Crossover Clinical Trial
Brief Title: Effect of Mediterranean Diet in Dyslipidemic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-Won Lee, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 3-2020-0030
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Dyslipidemias
Keywords: dyslipidemia; mediterranean diet; microbiome; inflammation; metabolic risk
MeSH Terms: conditions — Dyslipidemias; Inflammation | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet (Experimental): Mediterranean diet twice per day for four weeks
  Interventions: Behavioral: Mediterranean Diet
- Conventional diet (Placebo Comparator): Conventional diet for four weeks
  Interventions: Behavioral: Mediterranean Diet

INTERVENTIONS:
Behavioral: Mediterranean Diet — Diet instruction and menu samples from the dietitian on following the Mediterranean Diet.

SUMMARY:
The purpose of this randomized cross-over clinical trial is to examine the effects of Mediterranean diet based intervention on inflammation, metabolic risk and microbiome in patients with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* One or more of this criteria (total cholesterol ≥ 200mg/dl, LDL- cholesterol ≥130 mg/dL, triglyceride ≥ 200mg/dl)
* If woman of child bearing potential, agree to use effective contraception throughout the study period and 30 days after discontinuation of study drug
* Able to speak and read Korean
* Able to comply with all required study procedures and schedule
* Willing and able to give written informed consent
* Participants who are not participating in other clinical trials.

Exclusion Criteria:

* Participants with cancer treatment
* Participants with uncontrolled hypertension (systolic blood pressure (SBP) >180 mmHg, or diastolic blood pressure (DBP) >120 mmHg)
* Participants with uncontrolled diabetes or fasting glucose ≥ 200mg/dl)
* Participants with hepatic disease (aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >3 x institutional upper limit of normal) or renal disease (serum creatinine >2.0 mg/dL)
* Participants with significant cardiovascular disease (ischemic heart disease or stroke)
* Participants who are taking lipid-lowering medications.
* Participants who are taking other clinical trial medications.
* Participants with acute infectious disease such as pneumonia, acute gastroenteritis, and urinary tract infection.
* Vegetarian (does not eat red meat, poultry or fish)
* Participants with food allergy (sea food, fish, nuts, egg, meat, tomato, wheat, or soybean)
* Participants who are not able to eat more than 10 mediterranean meal in a row.
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | baseline, 4 weeks, 10 weeks
  body weight (kg)
Change in fat mass | baseline, 4 weeks, 10 weeks
  fat mass (kg) measured by bioelectrical impedance analyzer
Change in muscle mass | baseline, 4 weeks, 10 weeks
  muscle mass (kg) measured by bioelectrical impedance analyzer
Change in leukocyte count | baseline, 4 weeks, 10 weeks
  leukocyte count (/μL)
Change in C-reactive protein | baseline, 4 weeks, 10 weeks
  C-reactive protein (mg/L)
Change in fasting glucose | baseline, 4 weeks, 10 weeks
  fasting glucose (mg/dL)
Change in insulin | baseline, 4 weeks, 10 weeks
  insulin (mcIU/mL)

SECONDARY OUTCOMES:
Change in triglyceride | baseline, 4 weeks, 10 weeks
  triglyceride (mg/dL)
Change in high-density lipoprotein cholesterol (HDL-cholesterol) | baseline, 4 weeks, 10 weeks
  HDL-cholesterol (mg/dL)
Change in low-density lipoprotein cholesterol (LDL-cholesterol) | baseline, 4 weeks, 10 weeks
  LDL-cholesterol (mg/dL)
Change in gut microbiome | baseline, 4 weeks, 10 weeks
  Gut microbiome
Change in metabolomic response | baseline, 4 weeks, 10 weeks
  metabolomic profile of lipid metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Ji Won Lee, MD.PhD, Principal Investigator — Gangnam Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No